CLINICAL TRIAL: NCT05820854
Title: Patients' Self-care and Self-efficacy Scale in Oral Anticoagulation Therapy (SCSE-OAC): A Bilingual/Multi-national Mixed-method Validation Study
Brief Title: Self-care and Self-efficacy Scale in Oral Anticoagulation Therapy
Acronym: SCSE-OAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Arianna Magon, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: 164/INT/2022
Record Dates: First submitted 2023-04-05; First posted 2023-04-20 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Anticoagulants; Self Efficacy; Self Confidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-valvular atrial fibrillation (NVAF) patients treated with oral anticoagulants: Adult outpatients (≥ 18 years) with NVAF and treated with OAC for at least three months.
  Interventions: Other: Self-assess and reporting self-care self-efficacy levels

INTERVENTIONS:
Other: Self-assess and reporting self-care self-efficacy levels — Patients will have to self-report the self-care self-efficacy levels they experienced in managing the OAC therapy.

SUMMARY:
This study aims to develop and validate an index measurement tool to assess the patient's self-care self-efficacy in managing oral anticoagulation therapy (OAC). The index measure (i.e., SCSE-OAC) will be tested for its cross-cultural validity and reliability for the English and Italian-speaking population. For these reasons, a multi-phase and mixed-method observational and cross-sectional study design will be conducted.

DETAILED DESCRIPTION:
Oral anticoagulation therapy (OAC) is the most suitable treatment worldwide for the primary and secondary prevention of thromboembolism and stroke in patients with non-valvular atrial fibrillation (NVAF). However, the strategies to provide an optimal quality of anticoagulation control are still an open challenge for healthcare professionals. In this regard, understanding the health determinants underline the patient's adherence is fundamental in the research field to develop personalized patient-centered education interventions in clinical practice and consequently avoid low treatment adherence. Among these health determinants (e.g., patients' knowledge, health literacy, beliefs, etc), the patients' self-efficacy is underreported because a specific tool is not yet available to measure patients' self-efficacy regarding the health behaviors challenges in OAC self-care management.

The primary aim of this study is to develop the patients' self-care self-efficacy index in oral anticoagulation therapy management (SCSE-OAC) in adults with non-valvular atrial fibrillation and provide cross-cultural validity and reliability of the developed index measure.

More specifically, to assess the internal validity of the SCSE-OAC, content and construct validity proprieties will be tested for each translated version of the SECSE-OAC, as well as its reliability and invariance characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of non-valvular atrial fibrillation
* Outpatients
* Treating with any OAC for at least three months before enrollment
* Patients willing to participate in the study and provide informed consent

Exclusion Criteria:

* Patients treated with OAC for a brief period (i.e., less than three months)
* Patients with serious comorbidity (i.e, Charlson Comorbidity Index, ICC > 4)
* Patients who have suspended OAC for surgery in the last three months
* Cognitive impairment (assessed using six-item screener, SIS < 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each native-speaking country involved in the study will select a convenience sample of adult non-valvular atrial fibrillation patients (NVAF) chronically treated with oral anticoagulants.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
SCSE-OAC index | data collection will perform at the first 1 day patient visit
  The SCSE-OAC measurement index will provide evidence about the level patients perceive in their skills in facing daily challenges in managing their oral anticoagulation therapy. Furthermore, evidence of the validity and reliability of the SCSE-OAC tool will be provided for each native-speaking country involved in the study.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magon A, Hendriks J, Caruso R. Developing and Validating a Self-Care Self-Efficacy Scale for Oral Anticoagulation Therapy in Patients With Nonvalvular Atrial Fibrillation: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2024 Sep 13;13:e51489. doi: 10.2196/51489. PMID 39269742
- [Derived] Magon A, Hendriks JM, Conte G, Caruso R. Description of self-care behaviours in patients with non-valvular atrial fibrillation on oral anticoagulant therapy: a scoping review. Eur J Cardiovasc Nurs. 2024 Sep 5;23(6):582-591. doi: 10.1093/eurjcn/zvae007. PMID 38267024